CLINICAL TRIAL: NCT02508428
Title: A Prospective, Randomized Clinical Study Comparing Marathon Polyethylene and Enduron Polyethylene Acetabular Liners Used in Total Hip Arthroplasty at Long-Term Follow-up
Brief Title: Marathon and Enduron Polyethylene at Long-Term Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anderson Orthopaedic Research Institute (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AORI2015-0100
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Results first posted 2020-12-01 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases
Keywords: Osteolysis; Polyethylene; Crosslinked Polyethylene; Total Hip Replacement; Marathon
MeSH Terms: conditions — Osteoarthritis; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Osteolysis | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crosslinked Marathon polyethylene (Active Comparator): The crosslinked Marathon polyethylene liners used for the primary total hip replacements in this study were treated with 5 Mrad (50 kGy) of gamma irradiation to induce crosslinking and then heated above the melting temperature (150 degrees Celsius) to eliminate free radicals. This manufacturing process was designed to improve the polyethylene's resistance to wear through increased crosslinking and eliminate free radicals that render it susceptible to oxidative degradation. These liners were machined and terminally sterilized with gas plasma, a noncrosslinking chemical surface treatment. These liners did not have had free radicals at the time of implantation and did not incorporate antioxidants.
  Interventions: Device: Hip Replacement with crosslinked Marathon polyethylene
- Noncrosslinked Enduron polyethylene (Active Comparator): The standard, noncrosslinked Enduron polyethylene liners used for the primary total hip replacements in this study were manufactured from the same polyethylene resin as the crosslinked Marathon liners but never irradiated. Like the Marathon components, these liners were machined and terminally sterilized with gas plasma, a noncrosslinking chemical surface treatment. Based on the manufacturing methods, these liners would not have had free radicals at the time of implantation and did not incorporate antioxidants.
  Interventions: Device: Hip Replacement with noncrosslinked Enduron polyethylene

INTERVENTIONS:
Device: Hip Replacement with crosslinked Marathon polyethylene — Comparison of Marathon and Enduron polyethylene
  Arms: Crosslinked Marathon polyethylene
Device: Hip Replacement with noncrosslinked Enduron polyethylene
  Arms: Noncrosslinked Enduron polyethylene

SUMMARY:
The purpose of the study is to determine whether crosslinked Marathon and standard Enduron polyethylene liners show differences in survivorship due to wear-related revisions at minimum 14-year follow-up and every 5 years after.

DETAILED DESCRIPTION:
Several institutions have reported very low wear rates with crosslinked polyethylene based on early and midterm clinical data. However, since revisions associated with osteolysis typically occur after 10-year follow-up, the greatest benefits of the reduced wear associated with crosslinked polyethylene are expected to be reflected in lower revision rates for wear-related complications at long-term follow-up.

While crosslinking has proven to substantially reduce polyethylene wear during the first decade in vivo, characterizing the long-term clinical performance of Marathon polyethylene remains important because crosslinking is accompanied by a reduction in the ultimate tensile strength, fatigue strength, and elongation to failure of ultra high molecular weight polyethylene. As a consequence, concerns have been expressed about the potential for the liner fracture, in vivo polyethylene oxidation or accelerated wear at long-term follow-up, the effects of femoral head roughening over time and the bioreactivity of crosslinked polyethylene debris particles. Ultimately, the best way to address these concerns is in the context of well-controlled, long-term clinical outcome studies. This study will evaluate outcome at a minimum of 14-years after surgery among the same group of patients whose outcome was previously reported at 10-year follow-up. As part of our efforts to follow patients throughout their lives to obtain long-term outcome data, we will continue to obtain routine follow-up every 5 years from the date of the patient's primary total hip arthroplasty for the duration of the patient's life or until revision of the polyethylene liner (estimated to be 25 years). Because we anticipate that the reduced incidence of wear and osteolysis will result in a lower incidence of revision surgery among the patients randomized to Marathon liners, implant revision for reasons related to wear will be our primary outcome measure at long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

(from original study)

* Elective total hip replacement patient

(from 10-year follow-up)

* Consented to the original study.
* Received a Duraloc 100 cup with either a crosslinked Marathon or standard Enduron liner.
* Received an AML/Solution or a Prodigy stem with 28mm cobalt chrome femoral head.

Exclusion Criteria:

(from original study)

* None

(from 10-year follow-up)

* Patient did not receive device as specified in inclusion criteria.
* Patient refused to consent to continued follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 1999-01-06 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C. Anderson Engh, Jr., MD, Principal Investigator — Anderson Orthopaedic Research Institute
Locations (1):
- Anderson Orthopaedic Research Institute, Alexandria, Virginia, United States

REFERENCES:
- [Result] Leung SB, Egawa H, Stepniewski A, Beykirch S, Engh CA Jr, Engh CA Sr. Incidence and volume of pelvic osteolysis at early follow-up with highly cross-linked and noncross-linked polyethylene. J Arthroplasty. 2007 Sep;22(6 Suppl 2):134-9. doi: 10.1016/j.arth.2007.04.006. Epub 2007 Jul 27. PMID 17823032
- [Result] Engh CA Jr, Stepniewski AS, Ginn SD, Beykirch SE, Sychterz-Terefenko CJ, Hopper RH Jr, Engh CA. A randomized prospective evaluation of outcomes after total hip arthroplasty using cross-linked marathon and non-cross-linked Enduron polyethylene liners. J Arthroplasty. 2006 Sep;21(6 Suppl 2):17-25. doi: 10.1016/j.arth.2006.05.002. PMID 16950057
- [Result] Engh CA Jr, Hopper RH Jr, Huynh C, Ho H, Sritulanondha S, Engh CA Sr. A prospective, randomized study of cross-linked and non-cross-linked polyethylene for total hip arthroplasty at 10-year follow-up. J Arthroplasty. 2012 Sep;27(8 Suppl):2-7.e1. doi: 10.1016/j.arth.2012.03.048. Epub 2012 Jun 6. PMID 22682044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Beginning in January of 1999 and continuing over an 18-month period, patients at our institution were enrolled in a prospective, randomized, Institutional Review Board approved study to compare the outcome of THA using XLPE or CPE liners.
Pre-assignment Details: All patients undergoing primary THA were eligible to participate in this study. A total of 226 patients (236 hips) consented to participate. Six patients (6 hips) were excluded at the time of their surgery because they were not implanted with the study components for reasons related to intra-operative hip stability.
Units Other Than Participants: hips
Groups:
- Crosslinked Marathon Polyethylene: Total Hip Replacement using a crosslinked Marathon polyethylene liner
- Standard Enduron Polyethylene: Total Hip Replacement using a noncrosslinked Enduron polyethylene liner
Period: Overall Study
Arm/Group | Crosslinked Marathon Polyethylene | Standard Enduron Polyethylene
Started | 114; 116 hips | 111; 114 hips
Completed | 62; 64 hips | 44; 46 hips
Not Completed | 52; 52 hips | 67; 68 hips
Not completed — Death | 32 | 33
Not completed — Liner revised | 3 | 19
Not completed — Incomplete follow-up | 17 | 15

BASELINE CHARACTERISTICS:
Population: 230 hip replacements among 220 patients were randomized to crosslinked Marathon or noncrosslinked Enduron polyethylene liners.Among the 10 patients with bilateral hip replacements, two had both hips randomized to Marathon, three had both hips randomized to Enduron, and five had one hip randomized to Marathon and the other randomized to Enduron.
Units Other Than Participants: hips
Groups:
- Non-crosslinked Enduron Polyethylene: Total Hip Replacement using a noncrosslinked Enduron polyethylene liner
- Total: Total of all reporting groups
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene | Total
Number analyzed (Participants) | 114 | 111 | 220
Number analyzed (hips) | 116 | 114 | 230
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.6) | 62.0 (11.1) | 62.3 (10.8)
Sex: Female, Male [Count of Units; unit: hips]
  Female | 65 | 57 | 122
  Male | 51 | 57 | 108
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Weight [Mean (Standard Deviation); unit: pounds] | 186 (47) | 180 (40) | 183 (43)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter (kg/m^2)] | 28.6 (5.5) | 27.9 (5.1) | 28.2 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Hips Surviving at 15 Years
Description: Kaplan-Meier survivorship was calculated using revision for wear/osteolysis as an endpoint.
Time Frame: At 15-year follow-up and every 5 years after from the date of the patient's primary total hip arthroplasty for the duration of the patient's life or until revision of the polyethylene liner (estimated to be 25 years)
Population: All 230 total hip replacements randomized to crosslinked Marathon or non-crosslinked Enduron liners.
Measure: Number (95% Confidence Interval); unit: percentage of hips surviving at 15-years
Units Other Than Participants: hips
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene
Number analyzed (Participants) | 114 | 111
Number analyzed (hips) | 116 | 114
percentage of hips surviving at 15-years | 100 [100 to 100] | 86 [78 to 93]
Statistical Analysis 1: Comparison: Crosslinked Marathon Polyethylene vs Non-crosslinked Enduron Polyethylene; Survivorship was evaluated using liner revision for wear/osteolysis as an endpoint using a Kaplan-Meier analysis; Test type: Equivalence — Differences in survivorship among the Marathon and Enduron liners were evaluated with a Log Rank test; p < 0.001, Log Rank — A p-value of 0.05 was used as the threshold for statistical significance

2. Secondary Outcome: Polyethylene Wear
Description: A single reviewer, blinded to the type of polyethylene liner, evaluated femoral head penetration among all hips using serial anteroposterior pelvic radiographs. Two-dimensional head penetration was determined for each follow-up radiograph using Hip Suite Analysis version 8.0 with elliptical correction, a validated, computer-assisted technique. A linear wear rate was evaluated for each hip that had a minimum of three follow-up radiographs using a least-squares linear regression to calculate the slope of the best-fit line for the wear vector magnitude versus time in situ data. The slope from this regression represented the steady-state linear wear rate. The steady-state linear wear rate data from all hips in a group was used to compute a mean polyethylene wear value.
Time Frame: At minimum 14-year radiographic follow-up and every 5 years after from the date of the patient's primary total hip arthroplasty for the duration of the patient's life or until revision of the polyethylene liner (estimated to be 25 years)
Population: Hips with at least 3 serial anteroposterior pelvic radiographs that were revised or had minimum 14-year radiographic follow-up.
Measure: Mean (Standard Deviation); unit: mm/yr
Units Other Than Participants: hips
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene
Number analyzed (Participants) | 44 | 54
Number analyzed (hips) | 46 | 56
mm/yr | 0.03 (0.05) | 0.25 (0.16)
Statistical Analysis 1: Comparison: Crosslinked Marathon Polyethylene vs Non-crosslinked Enduron Polyethylene; Test type: Equivalence — Since the null hypothesis assumed that the wear rates were not different, "Equivalence" has been specified for the "Type of Statistical Test"; p < 0.001, t-test, 2 sided — A p-value of 0.05 was used as the threshold for statistical significance; Mean Difference (Net) = 0.22, 95% CI 2-sided [0.17 to 0.27]

3. Secondary Outcome: Incidence of Clinically Important Osteolysis Among Unrevised THAs
Description: The incidence of clinically important osteolysis is based on the number of unrevised THAs (total hip arthroplasties) with at least 1.5 square centimeters of pelvic and/or femoral osteolysis. Osteolysis was defined as an area of localized loss of trabecular bone or cortical erosion that was not apparent on the pre-operative or immediate postoperative radiograph. To obtain lesion sizes, the defects were outlined on the anteroposterior pelvic and lateral radiographs. The area of the osteolysis was measured using Martell's Hip Analysis Suite software. Lesions were considered clinically important if the total area of osteolysis around a hip replacement was at least 1.5 square centimeters on either the AP or lateral view.
Time Frame: as for outcome 2
Population: Unrevised hips that had minimum 14-year radiographic follow-up and revised hips that had a pre-revision radiograph available for analysis.
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene
Number analyzed (Participants) | 47 | 56
Number analyzed (hips) | 49 | 58
hips | 1 | 28
Statistical Analysis 1: Comparison: Crosslinked Marathon Polyethylene vs Non-crosslinked Enduron Polyethylene; Test type: Equivalence — Since the null hypothesis assumed that the incidences of clinically important osteolysis were not different, "Equivalence" has been specified for the "Type of Statistical Test"; p < 0.001, Fisher Exact — A p-value of 0.05 was used as the threshold for statistical significance; Risk Ratio (RR) = 0.04, 95% CI 2-sided [0.006 to 0.30]

4. Secondary Outcome: Patients Who Answered "Yes" to the Question, "Are You Satisfied With the Results of Your Hip Operation?"
Description: Patient satisfaction was quantified by asking participants to respond "yes" or "no" to the question, "Are you satisfied with the results of your hip operation?" Because some patients had both of their hips included in the study, these patients responded to the question, "Are you satisfied with the results of your hip operation?" for their right and left hips. As a consequence, the "Units Analyzed" is reported as hips while the "Number of Participants Analyzed" reflects the number of patients.
Time Frame: At minimum 14-year follow-up and every 5 years after from the date of the patient's primary total hip arthroplasty for the duration of the patient's life or until revision of the polyethylene liner (estimated to be 25 years)
Population: All patients with minimum 14-year follow-up who responded to the question, "Are you satisfied with the results of your hip operation?"
Measure: Count of Units; unit: hips
Units Other Than Participants: hips
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene
Number analyzed (Participants) | 51 | 47
Number analyzed (hips) | 53 | 49
hips | 53 | 48
Statistical Analysis 1: Comparison: Crosslinked Marathon Polyethylene vs Non-crosslinked Enduron Polyethylene; Since there were no patients with Marathon liners who were unsatisfied with the outcome of their hip replacement, a relative risk and the associated confidence interval could not be calculated; Test type: Equivalence — Since the null hypothesis assumed that the rate of satisfaction among the groups were not different, "Equivalence" has been specified for the "Type of Statistical Test"; p = 0.48, Fisher Exact — A p-value of 0.05 was used as the threshold for statistical significance

5. Secondary Outcome: Harris Hip Score
Description: The Harris Hip Score measures outcome after hip replacement and is based on a scale from 0 (worst) to 100 (best). The score includes assessments of pain, functional ability, deformity and range of motion.
Time Frame: as for outcome 4
Population: All hip replacements with minimum 14-year follow-up that had data to compute a Harris Hip Score.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Units Other Than Participants: hips
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene
Number analyzed (Participants) | 36 | 26
Number analyzed (hips) | 37 | 26
units on a scale | 96 [76 to 98] | 92 [74 to 95]
Statistical Analysis 1: Comparison: Crosslinked Marathon Polyethylene vs Non-crosslinked Enduron Polyethylene; Test type: Equivalence — Since the null hypothesis assumed that the Harris Hip Scores among the groups were not different, "Equivalence" has been specified for the "Type of Statistical Test"; p = .40, Wilcoxon (Mann-Whitney) — A p-value of 0.05 was used as the threshold for statistical significance

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from date of surgery up to 17 years after surgery.
Description: Reoperations were evaluated by reviewing medical records and asking patients if they had any additional surgery on their hip. Please note that adverse events are reported based on the number of hips enrolled in the study, not the number of patients. Ten patients had both of their hips included in the study including two who had both hips randomized to Marathon, three who had both hips randomized to Enduron and five who had one hip randomized to Marathon and the other randomized to Enduron.
Arm/Group | Crosslinked Marathon Polyethylene | Non-crosslinked Enduron Polyethylene
All-Cause Mortality (participants affected / at risk) | 32/116 | 33/114
Serious Adverse Events (participants affected / at risk) | 4/116 | 19/114
Other Adverse Events (participants affected / at risk) | 0/116 | 0/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crosslinked Marathon Polyethylene (N=116) | Non-crosslinked Enduron Polyethylene (N=114)
Wear/Osteolysis without fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (10) — Reopeartions for polyethylene wear and/or osteolysis without fracture of the bones around the hip joint
Recurrent Dislocation (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Wear/Osteolysis with Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) — Fractures included the greater trochanter, lesser trochanter and pubic ramus.
Open reduction of dislocation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The main weakness of this study is the incomplete followup. We attribute the incomplete followup to the unfortunate reality that older patients are frequently unwilling or unable to obtain followup for a variety of reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Materials should be submitted to the sponsor for review at least thirty days before they are due to be submitted for publication. The sponsor will inform the authors of any changes deemed necessary to preserve confidentiality, protect intellectual property or ensure scientific accuracy and the authors agree to make these changes before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT02508428/Prot_SAP_000.pdf